CLINICAL TRIAL: NCT01252056
Title: A Randomized, Control, Parallel, Open Label, Multi-centre Clinical Study to Evaluate the Efficacy and Safety of Cilostazol and Probucol in Combination on Patients With Diabetic Nephropathy
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Cilostazol and Probucol in Combination on Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260-09-805-01
Record Dates: First submitted 2010-04-21; First posted 2010-12-02 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Probucol; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Probucol (Active Comparator): Probucol treatment
  Interventions: Drug: Probucol
- Combination (Active Comparator): Probucol and Cilostazol
  Interventions: Drug: Probucol and Cilostazol

INTERVENTIONS:
Drug: Probucol — 250mg,Bid
  Arms: Probucol
Drug: Probucol and Cilostazol — 50-100mg,Bid
  Arms: Combination

SUMMARY:
The efficacy and safety of Cilostazol and Probucol in combination on patients with diabetic nephropathy is better than the single use.

DETAILED DESCRIPTION:
The objectives of this study is:

1. To evaluate the efficacy of Probucol on deferring nephropathy development of the patients with diabetic nephropathy (including: the change value of urine albumin from the baseline, the rate of the patients with serum creatinine reaching a doubling of the base-line serum creatinine, the rate of the hemodialysis-free survival).
2. To evaluate the efficacy of Cliostazol and Probucol in combination on deferring nephropathy development of the patients with diabetic nephropathy
3. To evaluate the efficacy of Cilostazol and Probucol in combination on atherosclerosis related biomarkers change. Atherosclerosis related biomarkers include:(a)Endothelium parameter: ICAM-1, vWF, VCAM-1,and McP-1. (b)Finolysis parameter: TM. (c)Inflammation parameter: Hs-CRP; IL-6. (d)Oxidation parameter: Ox-LDL, 8-OHdG. (e)Lipid parameter: TC, LDL-C, HDL-C, TG.
4. To evaluate the efficacy of Cilostazol and Probucol in combination on the progress of carotid intima-media thickness (IMT) on patients with diabetic nephropathy.
5. To evaluate the safety of Cilostazol and Probucol in combination on the patients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 40~75 years old
* Type 2 diabetes mellitus above 6 months
* HbA1c ≤8%
* Twice (above 2-week interval) confirmed urinary albumin at 30-3000µg/mg.cre
* Receive routine dosage ACEI or ARB treatment above 2 months, and the dosage has been fixed for at least 1 month
* LDL-C>100 mg/dL (2.60 mmol/L) and/ or hyperlipidemia patients with Statins treatment
* Free will to sign the informed consent form

Exclusion Criteria:

* Has an allergic history to investigational drugs
* Receive antilipemic agents (except Statins) within the latest 2 months, including Probucol
* Receive antiplatelet or anticoagulation agents (except Aspirin) within the latest 2 months, including Cilostazol
* Rapid progression of nephropathy within the latest 3 months
* Kidney disease caused by other reasons according to medical history
* Serum potassium level less than 3.5 mEq/L or more than 5.5 mEq/L
* Hemorrhagic tendency or hemorrhagic disease (such as alimentary tract hemorrhage, active fundus hemorrhage, etc.)
* Has a myocardial infarction, angina pectoris, or cerebral infarction within the latest 3 months
* Congestive heart failure
* Pregnant, potentially pregnant, or lactating woman
* Severe hepatic inadequacy (AST or ALT is 2.5 times higher than the upper limit of the normal value range)
* Serum creatinine level is 1.5 times higher than the upper limit of the normal value range
* Persistent or hardly controlled hypertension (such as malignant hypertension, SBP≥170 mmHg and/ or DBP≥100 mmHg)
* Severe ventricular arrhythmia (such as multiple and multifocal premature ventricular contractions)
* Has a medical history of cardiac syncope or primary syncope
* Has condition that may prolong QT interval (such as congenital long QT syndrome, taking drugs which prolong QT interval, hypokalemia or hypomagnesemia, etc.), or for man QT interval>450msec, for woman QT interval>470msec
* Has severe complication (such as diabetes mellitus ketoacidosis, nonketotic hyperosmolar diabetic coma, malignant tumor, severe anaemia, severe hematologic diseases, etc.)
* Register other clinical trials within the latest 3 months
* Other conditions that would be excluded from this study according to doctors'judgment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
nephropathy development | 96W
  After 96-week treatment, compare the efficacy between Probucol group and group control group on deferring nephropathy development of the patients with diabetic nephropathy (including: the change value of urine albumin from the baseline, the rate of the patients with serum creatinine reaching a doubling of the base-line serum creatinine, the rate of the hemodialysis-free survival)

SECONDARY OUTCOMES:
IMT | 48 and 96W
  After 48-week and 96-week treatment, compare the change value of IMT from the baseline among 3 modality groups.
Atherosclerosis related biomarkers | 48 and 96W
  After 12-week, 48-week and 96-week treatment, compare the change value of atherosclerosis related biomarkers from the baseline among 3 modality groups
Nephropathy development | 48 and 96W
  1. After 48-week and 96-week treatment, compare the efficacy among 3 modality groups on deferring nephropathy development of the patients with diabetic nephropathy (including: the change value of urine albumin from the baseline, the rate of the patients with serum creatinine reaching a doubling of the base-line serum creatinine, the rate of the hemodialysis-free survival)
Adverse events | 96W
  Incidence of adverse events, clinically relevant abnormal laboratory results before and after treatment (including hemotology, biochemistry, routine urine analysis and glycosylated hemoglobin), abnormal findings of vital sign, physical examination, and 12-lead ECG results

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Guo, Principal Investigator — Beijing University First Hospital
Locations (1):
- Beijing Universuty First Hospital, Beijng, Beijing Municipality, China

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730